CLINICAL TRIAL: NCT06499116
Title: Comparison of the Effectiveness of First-line Preventive Treatment of Migraine in Primary Care: a Pragmatic Clinical Trial [PREMI Study]
Brief Title: Comparison of the Effectiveness of First-line Preventive Treatment of Migraine in Primary Care
Acronym: PREMI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IJG-PREMI-2024; 2024-513597-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Migraine
Keywords: Migraine; Monthly Migraine Days (MMD); Preventive treatment; Primary care
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; Flunarizine; Amitriptyline; Propranolol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Topiramate (Experimental): 25-100 mg/12h, V.O., during 12 weeks
  Interventions: Drug: Topiramate
- Flunarizine (Experimental): 2,5-10 mg/24h, V.O., during 12 weeks
  Interventions: Drug: Flunarizine
- Amitriptyline (Experimental): 10-75 mg/24h, V.O., during 12 weeks
  Interventions: Drug: Amitriptyline
- Propranolol (Active Comparator): 20-120 mg/12h, V.O., during 12 weeks
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Topiramate — Treatment will be prescribed for GPs and they will decide the specific dosage 25-100 mg/12h.
  Other Names: Acomicil
  Arms: Topiramate
Drug: Flunarizine — Treatment will be prescribed for GPs and they will decide the specific dosage 2,5-10 mg mg/24h.
  Other Names: Sibelium
  Arms: Flunarizine
Drug: Amitriptyline — Treatment will be prescribed for GPs and they will decide the specific dosage 10-75 mg/24h.
  Other Names: Tryptizol
  Arms: Amitriptyline
Drug: Propranolol — Treatment will be prescribed for GPs and they will decide the specific dosage 20-120 mg/12h.
  Other Names: Sumial
  Arms: Propranolol

SUMMARY:
This study, which is aimed at comparing the effectiveness of the most frequently used drugs in the first line in primary care for the preventive treatment of migraine (amitriptyline, flunarizine, topiramate and propranolol), is a multicentre, pragmatic, parallel group, open randomised trial. Adults (≥18) candidates for preventive treatment for migraine; those with a frequency of ≥4 monthly migraine days, and who agree to participate in the clinical trial, will be randomised to one of the 4 groups. Sample: 460 patients. The primary outcome will be the reduction in monthly migraine days, comparing amitriptyline, flunarizine and topiramate with propranolol.

ELIGIBILITY:
Inclusion Criteria:

- Adults (≥18) candidates for preventive treatment for migraine; those with a frequency of ≥4 monthly migraine days, and who agree to participate in the clinical trial.

Exclusion Criteria:

* People diagnosed with migraine who are not candidates for preventive migraine treatment
* People diagnosed with chronic migraine (>15 days of headache per month, of which 8 are monthly migraine days)
* Not having a smartphone
* Simultaneous participation in another clinical trial
* Pregnancy or expected pregnancy during the next 3 months
* Lactation
* People with migraine who already receive preventive treatment.
* People on chronic treatment with opioids or other analgesics or NSAIDs that are not used for the symptomatic treatment of migraine, for example, osteoarthritis.
* People who, in the opinion of the clinician, have an absolute contraindication to one of the study drugs or who cannot perform the trial procedures:

Hypersensitivity to any of the study drugs / Heart block or severe bradycardia / Concomitant treatment with verapamil or diltiazem / Active cardiovascular pathology (recent heart attack, angina, Raynaud's phenomenon) / Major depression or active treatment with antidepressants (including monoamine oxidase inhibitors and St. John's wort) / Other psychiatric illnesses or active treatment with antipsychotics or lithium / Severe liver disease or kidney failure / Parkinson's disease or other extrapyramidal disorders / Epilepsy (diagnosis and/or active treatment) / Any other contraindication that, in the opinion of the clinician, prevents participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the most frequently used drugs in primary care for the preventive treatment of migraine according to the reduction in monthly migraine days, comparing amitriptyline, flunarizine and topiramate with propranolol. | 12 weeks
  Clinical effectiveness: change in the mean number of monthly migraine days (MMD) at 12 weeks of treatment from baseline.

SECONDARY OUTCOMES:
Calculate the rate of responders (reduction of at least 50% in monthly migraine days compared to baseline) | 12 weeks
  Proportion of patients responding at 12 weeks from start of treatment; <25% change in mean number of MMD: non-responders, 25-49%: partial responders, 50-75%: responders, >75%: excellent responders.
Evaluate effectiveness before completing the clinical trial | 4, 8 and 12 weeks
  Change in mean number of MMDs at 4 and 8 weeks from baseline.
Estimate the reduction in the intensity of migraine attacks | 4, 8 and 12 weeks
  Reduction in the mean number of moderate-severe MMD at 4, 8 and 12 weeks from the start of treatment.
Estimate the prevalence of symptoms associated with migraine | 12 weeks
  Proportion of patients with associated symptoms at 12 weeks from the start of treatment; photophobia, phonophobia, nausea.
Evaluate adherence to preventive treatment | 12 weeks
  Proportion of adherent and non-adherent patients (according to taking [yes/no] of the study treatment with the prescribed dosage) at 12 weeks from the start of treatment.
Estimate the reduction in the use of symptomatic treatment drugs used to treat migraine attacks (analgesics, NSAIDs, triptans, others). | 4, 8 and 12 weeks
  Change in the mean number of drugs used for symptomatic treatment at 4, 8 and 12 weeks from baseline.
Evaluate reconsultation visits due to migraine attacks | 4, 8 and 12 weeks
  Reconsultations: Type of consultation (PCC, PC emergency, hospital, hospital emergency). Number of consultations after 12 weeks from the start. Number of medical tests performed relacionadas con la migraña.
Evaluate improvement in quality of life and patient satisfaction | 12 weeks
  Change in EQ-5D-5L questionnaire at 12 weeks from baseline. Including Visual Analogue Scale (0-100). Lower scores means worse health condition.
Analyze the differences between men and women regarding study drugs effectiveness. | 4, 8 and 12 weeks
  Result comparison change in mean number of MMDs adjusted by sex
Estimate the disability associated with migraine attacks according to number of paticipans reporting temporary work disability, absenteeism, presenteeism. | 12 weeks
  Change in the number of ILT days, absenteeism, presenteeism at 12 weeks from the start of treatment.
Incidence of adverse events of the four drugs used in the preventive treatment of migraine . | 12 weeks
  Number of adverse events

IPD SHARING:
Plan to Share IPD: No
All publications will be free and open access. Publications of clinical trial results are planned in national and/or international scientific journals and in communications to conferences. Results will also be communicated to scientific societies and other actors involved in decision-making in the healthcare field, as well as through dissemination activities to patients and citizens in general.

REFERENCES:
- [Derived] Giner-Soriano M, Morros R, Monfa R, Ouchi D, Fernandez-Garcia S, Vedia C, Bonet Monne S, Calvo Martinez EM, Copetti Fanlo S, Morollon N, Belvis Nieto R, Delgado-Espinoza CE, Garcia-Sangenis A. Comparison of the effectiveness of first-line preventive treatment of migraine in primary care: study protocol for a pragmatic clinical trial (PREMI study). Trials. 2025 Aug 26;26(1):311. doi: 10.1186/s13063-025-08961-0. PMID 40859286